CLINICAL TRIAL: NCT07139496
Title: Combined Injury-site & Lumbosacral Epidural Stimulation for Spinal Cord Injury - a Pilot Study.
Brief Title: Combined Injury-site & Lumbosacral Epidural Spinal Cord Stimulation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Chan Chi-Wing, Consultant, Department of Anaesthesia, Pain & Perioperative Medicine, The University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UW 25-294
Record Dates: First submitted 2025-07-07; First posted 2025-08-24 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Spinal Cord Injuries (SCI)
Keywords: Injury-site; Lumbosacral Epidural Stimulation; Spinal Cord Injury; Spinal cord stimulation
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Spinal Cord Stimulator (Experimental): After signing the consent form, the patient will be assigned for standard surgery with additional implant of the spinal cord stimulator. Two percutaneous SCS leads will be placed at the level of SCI. These leads were anchored and were tunneled to subcutaneous space in posterior iliac crest and were connected to impulse generator. Another two percutaneous SCS leads will be placed over the lumbrosacral spinal cord. Intraoperative neurological monitoring will be performed. The aim is to determine spinal segmental mapping and to elicit evoked action potentials with contraction of muscles related to locomotor function of the lower limbs. These leads were anchored and were tunneled to subcutaneous space in posterior iliac crest and were connected to impulse generator.
  Interventions: Device: Spinal Cord Stimulator

INTERVENTIONS:
Device: Spinal Cord Stimulator — After the implantation of the spinal cord stimulator, the study will begin with 3 phases:
  For the first phase, SCS over lumbrosacral spinal cord will be activated for 3 months with appropriate stimulation of lower limb muscles for walking.
  For the second phase, SCS over lumbrosacral spinal cord will be stopped. SCS over the injury site will be activated for 3 months with appropriate stimulation of lower limb muscles for walking.
  For the third phase, SCS over both lumbrosacral spinal cord and injury site of spinal cord will be activated for another 3 months with appropriate stimulation of lower limb muscles for walking
  During all the phrases, physiotherapy of individual muscle groups for walking will be arranged. Exoskeleton training will also be arranged for 4 to 5 hours per week.

SUMMARY:
Spinal cord stimulation (SCS) has been shown in previous studies to be capable of restoring motor and autonomic function in patients with chronic complete spinal cord injury (SCI). Clinical studies have demonstrated that SCS enables activation of previously paralyzed muscles, leading to functional improvements in patients in the chronic stage of paralysis through the delivery of activity-based interventions. For most previous studies on SCS in SCI, stimulation was invariably applied to lumbrosacral plexus only. In this study, after signing the consent form, the patient will be assigned for standard surgery with additional implant of the spinal cord stimulator. The investigators propose to conduct the SCS with three phases. For the first phase, SCS over lumbrosacral spinal cord will be activated for 3 months with appropriate stimulation of lower limb muscles for walking together with physiotherapy of individual muscle groups for walking. For the second phase, SCS over lumbrosacral spinal cord will be stopped. SCS over the injury site will be activated for 3 months with appropriate stimulation of lower limb muscles. For the third phase, SCS over both lumbrosacral spinal cord and injury site of spinal cord will be activated for another 3 months with appropriate stimulation of lower limb muscles.

DETAILED DESCRIPTION:
Spinal cord injury (SCI) causes damage to motor, sensory, and autonomic function below the level of injury. This can have a huge impact on the daily function of the patients, with devastating effects on their quality of life, especially those with paralysis. Surgical treatment including decompression surgery is an option to improve the neurological outcome of these patients if the paralysis or limb weakness were surgically correctable. However, even with surgical treatment, there are still many patients with residual neurological deficits, which may greatly impair their activities of daily living. Patients with post-SCI may also develop chronic debilitating pain, because of neurophysiological changes in the somatosensory system.

Spinal cord stimulation (SCS) has increasingly been used as a potential method of improving motor function and for pain relief in patients with spinal cord injury. SCS is a well-established therapeutic treatment with robust evidence, in the management of chronic neuropathic and ischaemic pain syndromes, including persistent back pain after surgery, complex regional pain syndrome, and chronic ischemic pain condition. Its proposed mechanism of analgesic effects includes the gate control theory of pain, and enhancement of GABAergic systems of dorsal horn cells by stimulating their dendrites. Currently, there is a lack of mechanistic studies of SCS for SCI pain and its effectiveness is not well established.

SCS has been shown in previous studies to be capable of restoring motor and autonomic function in patients with chronic complete spinal cord injury. Clinical studies have demonstrated that SCS enables activation of previously paralyzed muscles, leading to functional improvements in patients in the chronic stage of paralysis through the delivery of activity-based interventions. For most previous studies on SCS in SCI, stimulation was invariably applied to lumbrosacral plexus only. The proposed mechanism for the effects of relate to the increased excitability of the central pattern generators (CPG) and enhance tonic and rhythmic motor patterns in persons after SCI and results in the activation of lower extremity muscles for standing and stepping with and without assistive devices. It was also shown that SCS in combination with locomotor training provides sensorimotor training of the spinal circuitry and facilitates standing stepping to enhance neuroplasticity.

In this study the investigators hypothesize that the application of SCS to the injury site can provide a neuromodulatory effect to the recovering neurons, allowing for improved neurological function caudal to the injury site. The investigators propose to conduct a clinical trial to determine whether the application of SCS to both injury site and lumbrosacral spinal cord, instead of SCS over lumbrosacral spinal cord alone, can further improve motor function in patients with motor-complete subacute and chronic spinal cord injury. The investigators will also assess longer term secondary outcomes including lower limb functional scores, chronic pain, and health related quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. American Society of Anesthesiologist (ASA) status I-III
2. Age 18-70 years old
3. Patients with SCI more than 2 years
4. Traumatic or atraumatic spinal cord injury
5. American Spinal Injury Association (ASIA) Impairment Scale A and B
6. Have previous MRI to document extent of spinal cord injury before recruitment

Exclusion Criteria:

1. Chronic opioid user
2. Presence of chronic pain condition (pain duration over 3 months)
3. Alcohol or substance abuse
4. active and unaddressed psychiatric diseases

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2028-09-01 (Estimated); Study Completion 2029-03-01 (Estimated)

PRIMARY OUTCOMES:
Assisted/independent standing or stepping (A/I) [Time Frame: Changes from baseline to the third phase of the intervention] | From baseline to three months after the third phase of the intervention.
  Assisted/independent standing or stepping of participants will be recorded, with 0 = unable, 1 = maximal assistance, 2 = moderate assistance, 3 = independent with device, 4 = fully independent.
Gait analysis (GA) [Time Frame: Changes from baseline to the third phase of the intervention] | From baseline to three months after the third phase of the intervention.
  The participants' hip, knee range of motion will be recorded. The walking speed will also be recorded.
Overground walking (OGW) [Time Frame: Changes from baseline to the third phase of the intervention] | From baseline to three months after the third phase of the intervention.
  The speed, time and distance for the participants' overground walking will be recorded.
Treadmill stepping/ walking (TSW) [Time Frame: Changes from baseline to the third phase of the intervention] | From baseline to three months after the third phase of the intervention.
  The maximum tolerated speed (m/s) and duration (minutes) for treadmill stepping/walking will be recorded.
Walking Index for Spinal Cord Injury Scale (WISCI 2) [Time Frame: Changes from baseline to the third phase of the intervention] | From baseline to three months after the third phase of the intervention.
  A score from 0 to 20 will be recorded for WISCI II. Level 0: "patient is unable to stand and/or participate in assisted walking" to level 20: "ambulates with no devices, no braces and no physical assistance, 10 meters".
Sensory assessments of the lower limbs [Time Frame: Changes from baseline to the third phase of the intervention] | From baseline to three months after the third phase of the intervention.
  The sensory changes of the participants will be recorded with 'absent', reduced' or 'present'.

SECONDARY OUTCOMES:
Pain Intensity [Time Frame: Changes from baseline to the third phase of the intervention] | From baseline to three months after the third phase of the intervention.
  NRS pain scores with movement will be recorded (NRS scale 0-10, where 0 is no pain, and 10 is the worst possible pain)
Quality of Life [Time Frame: Changes from baseline to the third phase of the intervention] | From baseline to three months after the third phase of the intervention.
  A SF36 questionnaire with scores range from 0 to 100 for eight domains will be recorded, with a higher score defining a more favorable health state. The eight domains include: physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue, and general health perceptions.
Psychological Symptoms [Time Frame: Changes from baseline to the third phase of the intervention] | From baseline to three months after the third phase of the intervention.
  The Depression and Anxiety Symptom Stress Scale (DASS) of participants will be recorded. A score range from 0 to 42 in depression, anxiety and stress will be recorded with a higher score meaning a more severe psychological symptom.
Presence of neuropathic pain [Time Frame: Changes from baseline to the third phase of the intervention] | From baseline to three months after the third phase of the intervention.
  A score of 3 or higher from an Identification Pain Questionnaire will be used to indicate the likely presence of neuropathic pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Queen Mary Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No